CLINICAL TRIAL: NCT05787626
Title: Efficacy of the Transverse Planes Technique in the Diaphragmatic Region in Young Subjects. A Randomized Controlled Trial
Brief Title: Efficacy of the Transverse Planes Technique in the Diaphragmatic Region in Young Subjects.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidad Católica San Antonio de Murcia (Other)
Responsible Party: Principal Investigator, Jasemin Todri, Principal Investigator, Universidad Católica San Antonio de Murcia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CE022305
Record Dates: First submitted 2023-03-03; First posted 2023-03-28 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Healthy; Diaphragm Issues

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional group (Experimental): The intervention consists of the application of a myofascial technique in the diaphragmatic region, one hand of the therapist will be placed on the hemidiaphragm to be treated and the other hand on the same side but on the dorsal part of the patient on the costal edge of the last ribs.
  Interventions: Other: manipulation
- Control group (Sham Comparator): In the subjects of the control group, the hands will be placed in the same position but without any therapeutic intention, applying the minimum possible pressure.
  Interventions: Other: manipulation

INTERVENTIONS:
Other: manipulation — miofascial technique in diaphragmatic region

SUMMARY:
In the present study, 28 healthy young people will be selected, who will be evaluated by a blind investigator regarding the study objectives, and will be randomly included in two groups. The experimental group will consist of 14 subjects who will carry out 1 weekly session of 10 minutes and who will be evaluated just before starting the intervention, after it and at 4 weeks. The control group will be made up of 14 subjects who will be evaluated in the three periods described without the need to carry out the intervention.

DETAILED DESCRIPTION:
The intervention will be carried out for 4 weeks, with 1 weekly session of 10 minutes duration. The patient will go to the intervention room where the treatment procedure will be explained in detail. He will be explained verbally and with a visual demonstration of what the technique consists of and how it is going to be performed, the position that he has to adopt during and how long the intervention will last.

The intervention consists of the application of a myofascial technique in the diaphragmatic region, one hand of the therapist will be placed on the hemidiaphragm to be treated and the other hand on the same side but on the dorsal part of the patient on the costal edge of the last ribs.

The patient will be asked to focus on their own breathing and the contact that the therapist will apply.

In the subjects of the control group, the hands will be placed in the same position but without any therapeutic intention, applying the minimum possible pressure.

ELIGIBILITY:
Inclusion Criteria:

* Healthy people
* no spinal pathology
* no respiratory pathology

Exclusion Criteria:

* have suffered spinal pathologies in the last 3 months
* have suffered respiratory diseases in the last 3 months

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Estimated)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2023-05-01 (Estimated); Study Completion 2023-05-30 (Estimated)

PRIMARY OUTCOMES:
Centimetric measurement of the thorax | change from baseline to one month
  measuring the difference in circumference after maximum inhalation through the nose and maximum exhalation through the mouth, the measurement is made at the level of the xiphoid process
Back range of motion | change from baseline to one month
  Performing the Ott Test, which consists of performing, with the subject standing, two measurements, one in the lower part of the spinous process of C7 and the other 30 centimeters below the previous mark.
Inspiratory and expiratory capacity | change from baseline to one month
  will be carried out using an incentive spirometer